CLINICAL TRIAL: NCT06762574
Title: "Effect of Low Level Laser Therapy on Neuropathic Pain After Neck Dissection Surgery''
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dalia Fathi Ragab Gawish, Physical therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Neck dissection surgery
Record Dates: First submitted 2024-12-23; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Neck Disease, Head and Neck Cancer; Neuropathic Pain
Keywords: Neck dissection surgery; Neuropathic pain; Rang of motion
MeSH Terms: conditions — Head and Neck Neoplasms; Neuralgia | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group receive low level laser Therapy and traditional medical treatment (Active Comparator)
  Interventions: Other: Low Level Laser Therapy
- Control group receive placebo Low Level Laser Therapy and traditional medical treatment (Placebo Comparator)
  Interventions: Other: Placebo Low Level Laser Therapy

INTERVENTIONS:
Other: Low Level Laser Therapy — Low Level Laser Therapy sometimes known as Low Level Light Therapy or Photobiomodulation (PBM) is a low intensity light therapy. The effect is photochemical not thermal. The light triggers biochemical changes within cells and can be compared to the process of photosynthesis in plants, where the photons are absorbed by cellular photoreceptors and triggers chemical changes.
  Arms: Study group receive low level laser Therapy and traditional medical treatment
Other: Placebo Low Level Laser Therapy — Placebo Low Level Laser Therapy:turning on the device with covering probe by aluminum foil and ask patient to wear sun glasses to obtain the placebo effect.
  Arms: Control group receive placebo Low Level Laser Therapy and traditional medical treatment

SUMMARY:
The purpose of the study was to evaluate the effect of Low Level Laser Therapy on neuropathic pain after neck dissection surgery.

It was hypothesized that: Low Level Laser Therapy is effective on improving Neuropathic pain post neck dissection surgery .

DETAILED DESCRIPTION:
Patients diagnosed with head and neck cancer are treated with surgery, radiation therapy and/or chemotherapy, with the aim of maximizing survival whilst preserving physical form and function .The surgical dissection of the neck is a typical technique for the management of head and neck malignant growths from the squamous cell carcinoma .

Neck dissection (ND) is performed for known metastatic neck disease, prophylactically in cases where there is increased risk for occult metastatic disease or as a staging procedure. Neck dissection (ND) is used to treat known metastatic neck disease, as a preventative measure against occult metastatic disease. A common surgery for treating malignant growths of the head and neck caused by SCC is surgical ND.

There are various approaches to performing the neck dissection surgery. One of these approaches is the radical neck dissection that involves the total excision of lymph nodes from one side of the neck, the muscle that helps turn the head (sternocleidomastoid muscle), a significant vein (internal jugular vein), and a nerve that is essential in the full-range of movement of the arm and shoulder (spinal accessory nerve).In contrast, the modified radical neck dissection preserves one or more of the aforementioned important structures .

Neck morbidity was common and apparent after cancer treatment; this includes limited ROM, impairment of sensations, and neck pain . In an investigation of 25 patients with permanent neck pain following neck dissection, two types of neck pain were described;neuropathic and myofascial pains.

Furthermore, shoulder and neck symptoms were reported in 37% and 33% of 220 participants who had neck dissection surgery , respectively, while myofascial and neuropathic pains were reported in 46% and 32% of the patients, respectively .

A new definition of pain has been formalized and adopted by International Association for the Study of Pain in January 2020, which states that pain is "An unpleasant sensory and emotional experience associated with or resembling that associated with actual or potential tissue damage".

Surgical resection of a tumor is associated with intractable pain of the shoulder, neck, and craniofacial areas. Correct identification of structures such as the cervical plexus and the spinal accessory nerve reduces the manifestation of chronic pain states . Parwis Agha-Mir-Salim et al. showed the essential role played by the cervical plexus in the development of chronic pain with neuropathic characteristics after several types of radical neck dissections. The cervical plexus is essential for sensory innervation of the cervical region and the skin of the shoulder. It is formed by the anterior division of the first four cervical nerves and it is a sensory anatomical substrate for this region .

Damage of the cervical rootlets during neck dissection may lead to neck sensory abnormality (anesthesia, numbness, and/or neuropathic pain), edema and limitation of neck/shoulder movement, decline in speech and eating abilities.

Neuropathic pain is usually managed with a variety of pharmacological and non-pharmacological therapies Among nonpharmacological treatments Transcranial Electrical Stimulation , acupuncture, massage therapy and Transcutaneous .Recent studies have reported the use of laser therapy in patients with peripheral somatosensory neuropathy and neuropathic pain .Specifically, clinical studies on the effects of laser therapy on injured nerve reported an increase in nerve function .

ELIGIBILITY:
Inclusion Criteria:

* Fiftyـtwo patients of both genders with age ranged between 30 to 60 years will participate in this study.
* All patients had neuropathic pain following Unilateral radical neck dissection surgery.
* All patients had history of neuropathic pain involving superficial cervical plexus after unilateral radical neck dissection surgery.
* All patients had moderate or severe pain of tingling,numbness and electric nature following neck dissection surgery. NP confined to the C2-C4 distributions, involves one or more branches of the SCP;especially in the skin overlying lateral neck .
* Informed consent was obtained from every patient enrolled in the trial.
* Moderate to severe pain (VAS score >4).

Exclusion Criteria:

* A wound in the affected area.
* A cervical disk lesion.
* Cervical spine fracture or spondylolisthesis.
* Rheumatoid arthritis.
* Epilepsy or any psychological

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-01-06 (Estimated); Primary Completion 2025-01-13 (Estimated); Study Completion 2025-02-13 (Estimated)

PRIMARY OUTCOMES:
Neck Neuropathic pain | 6 weeks
  * Douleur Neuropathique 4 questionnaire : It is a screening questionnaire to identify neuropathic pain in clinical practice and research, it showed significant accuracy of 83% sensitivity and 90% specificity.It is made up of seven items related to symptoms and three items related to physical evaluation . Each item is scored 1 if the answer is positive and zero if negative, leading to a minimum score of zero and maximum of 10. Cut-off point is four, being that scores equal to or above 4 suggest neuropathic pain .

SECONDARY OUTCOMES:
Neck pain | 6 weeks
  *Visual analogue scale :for acute pain measurement. is the most widely used technique for assessing pain intensity , a continuous scale with a vertical or horizontal line of 100 mm, from 0 to10, whose extremes are designated "no pain" and "worst imaginable pain" (0= no pain; 10= most painful imaginable pain). Patients were instructed to indicate how severe the pain was on that line
Neck Rang of motion | 6 weeks
  *Goniometer: is a reliable method to evaluate active Rang of motion clinically.
  ROM of the cervical spine is approximately:
  80° to 90° of flexion, 70° of extension, 20° to 45° of lateral flexion, Up to 90° of rotation to both sides.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] de Pedro M, Lopez-Pintor RM, de la Hoz-Aizpurua JL, Casanas E, Hernandez G. Efficacy of Low-Level Laser Therapy for the Therapeutic Management of Neuropathic Orofacial Pain: A Systematic Review. J Oral Facial Pain Headache. 2020 Winter;34(1):13-30. doi: 10.11607/ofph.2310. Epub 2019 Jul 24. PMID 31339967
- [Background] de Andrade AL, Bossini PS, Parizotto NA. Use of low level laser therapy to control neuropathic pain: A systematic review. J Photochem Photobiol B. 2016 Nov;164:36-42. doi: 10.1016/j.jphotobiol.2016.08.025. Epub 2016 Aug 31. PMID 27639607